CLINICAL TRIAL: NCT06534151
Title: Virtual Twins and Tools for Personalised Clinical Care- the Heart Failure With Reduced Ejection Fraction Sub-study
Brief Title: VITAL - the Heart Failure With Reduced Ejection Fraction Sub-study
Status: Not yet recruiting | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 173420
Record Dates: First submitted 2024-07-19; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Heart failure with reduced ejection fraction; Cardiac resynchronisation therapy; Digital twin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will undergo immediate laboratory testing for haematocrit and renal function (point of care testing).
  Other blood samples and a urine sample will be stored for later proteomics (including where applicable metabolomics and lipidomics and other small molecule analysis) and gene code analysis (DNA/RNA). The investigators may look at all or part of the DNA code, even if it has been looked at before, and at the RNA code (RNA is the version of the DNA code that the body uses to make proteins).
  Blood cells will be collected for future derivation of human pluripotent cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing implantation of cardiac resynchronisation therapy (CRT) device: These patients will have a diagnosis of heart failure with reduced ejection fraction (confirmed by a heart scan called an echocardiogram). A consultant cardiologist will advise they have a CRT device implanted to improve their symptoms and quality of life.
  Interventions: Device: CRT implantation

INTERVENTIONS:
Device: CRT implantation — A CRT is a device (that looks like a pacemaker) that will be used to help the ventricles contract synchronously.

SUMMARY:
Heart failure affects over 1 million people in the United Kingdom. Approximately 50% have heart failure with reduced ejection fraction (HFrEF), a condition where the heart muscle does not contract properly. If the right and left chambers (called 'ventricles') of the heart are not pumping at the same time, devices called cardiac resynchronisation therapy (CRT) can be inserted to encourage the ventricles to pump together, reducing heart failure symptoms and helping people to live longer.

CRT devices are made of wires which are placed into the ventricles through the blood vessels that carry blood to and from the heart. However, one third of patients do not show any improvement following CRT insertion, and another third show only a partial improvement. Doctors cannot accurately predict who will respond well, meaning patients may undergo a procedure with no benefit, being exposed to risks including bleeding and infection.

Virtual models of a patient's heart and blood vessels, known as a 'digital twin', can be generated using artificial intelligence. These models can be used to predict a patient's response to a procedure without them having to undergo the procedure first, meaning patients can avoid being exposed to risks.

30 patients with HFrEF who have been selected to have CRT implanted by their consultant cardiologist will be recruited. Before having their procedure patients will attend University College London (UCL) for tests including a blood test, urine test, magnetic resonance imaging (MRI) scan of the heart, ultrasound of the heart, a 5-minute heart recording and a 6- minute walking/ stepping test. After the CRT is implanted, the patient's response to the device will be assessed with a blood test, a 6-minute walking/ stepping test and a heart ultrasound scan 3 and 6 months after the procedure. The virtual models will be used to determine if a patient's response to CRT can be accurately predicted.

DETAILED DESCRIPTION:
Heart failure affects over 1 million people in the United Kingdom. Approximately 50% of these people have heart failure with reduced ejection fraction (HFrEF), a condition where the muscle of the heart does not contract properly. Without treatment, patients are at risk of developing fluid around the lungs and legs (called oedema), abnormal heart rhythms (known as arrhythmias), and death. Treatment involves a combination of tablets, but some patients show no improvement with medications. When the left and right chambers of the heart are not pumping at the same time, devices called cardiac resynchronisation therapy (CRT) can be implanted to encourage the chambers to pump together, reducing symptoms and improving the patient's quality of life.

CRT devices consist of wires which are placed into the ventricles through the blood vessels which lead to the heart. However, despite an initially successful procedure, over one third of patients do not show any improvement following CRT implantation. Risks associated with the procedure include bleeding, infection and damage to the underlying lung or heart muscle (which can be life-threatening), meaning a significant proportion of patients undertake these risks with no benefit afterwards. Moreover, the infection risk is lifelong, and patients may develop device-related infective endocarditis at any stage, which is associated with a high mortality.

Virtual models of a patient's anatomy and blood flow, known as a 'digital twin', can be generated using artificial intelligence. These models can be used to predict a patient's response to a treatment or procedure. Digital twins have been studied in research projects looking at coronavirus disease 2019 (COVID-19), asthma and cancer. Within cardiology, digital twins have been studied in patients who are undergo valve surgery. So far, no models have been developed to predict patients' responses to heart failure treatments.

Working closely with bioengineers, physiologists and computer scientists, this study aims to develop a validated, multi-scale, multi-organ modelling platform than can create an individualised virtual twin, incorporating cardiovascular anatomy as well as complex physiological processes including the inter-connection of organ systems, the autonomic nervous system activity and hormonal actions.

A minimum of 30 patients who are undergoing a clinically-indicated implantation of CRT will be recruited. Before the procedure, each patient will attend University College London (UCL) for a range of tests including measurement of height, weight and blood pressure, an echocardiogram, a cardiac magnetic resonance imaging (MRI) scan, a 12-lead electrocardiogram (ECG), a 256-lead electrocardiographic imaging recording (a 5-minute detailed recording of the heartbeat), a 6-minute walking/ stepping test and blood and urine sample collection. A subset of patients will also be provided with a wearable heart monitor which will be worn during their UCL appointment. These data will be integrated into the modelling framework to create a personalised virtual 'twin' for each patient.

Following implantation of the CRT, each patient will return for follow-up visits at 3 months and 6 months when they will undergo a further echocardiogram, blood test and 6 minute step/walk test.

A clinically-validated virtual platform would have the potential to transform how patients are selected to undergo device implantation in the following ways:

* Patients who are predicted to be 'non-responders' can be directed to other treatments and avoid the serious potential risks associated with device implantation.
* Device selection can be optimised. There are 2 forms of CRT:

  1. Biventricular pacing (BiVP) which involves implanting one lead into each ventricle
  2. Conduction system pacing (CSP) which requires placement of a lead into the conducting heart tissue in the septum between the ventricles.

CSP is considered to better mimic the heart's own physiology, but is more technically challenging to achieve, often leading to a longer and higher risk procedure. Patients referred for both forms of CRT will be recruited to this study. A validated modelling platform may be able to predict which form of pacing would benefit the patient most, meaning clinicians will be able to select the optimal form of pacing without exposing a patient to unnecessary complications.

ELIGIBILITY:
Inclusion Criteria:

* Age: >18 years old
* Confirmed indication for CRT-device implantation (heart failure with reduced ejection fraction and dyssynchrony on ECG)

Exclusion criteria:

* Pregnancy
* Any typical contra-indication to a MRI scan (e.g. ferromagnetic fragments in the body
* Chronic kidney disease stage 4 or 5)
* Not able to mobilise (as they will not be able to participate in a 6 minute step test)
* Extreme frailty or life expectancy < 6 months
* Recent myocardial infarction within 3 months
* Cardiac revascularisation or valve surgery/ implantation within the last 3 months
* Participation in a trial that includes active treatment
* Anyone with untreated symptomatic cardiovascular disease or severe hypertension

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will a known diagnosis of heart failure with reduced ejection fraction (seen on echocardiogram) and ventricular dyssynchrony (seen on ECG) who are symptomatic despite medical treatment, so meet criteria to have a CRT device fitted as per guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Ejection fraction measured by 3-dimensional echocardiography | 3 months
  An ultrasound of the heart that measures how well the heart muscle is contracting.
6-minute step/walk test | 3 months
  An assessment of how may steps a patient can take in 6 minutes
6-minute step test | 6 months
  An assessment of how may steps a patient can take in 6 minutes
Ejection fraction measured by 3-dimensional echocardiography | 6 months
  An ultrasound of the heart that measures how well the heart muscle is contracting.
Blood test | 6 months
  Blood test to measure N-terminal pro-brain natriuretic peptide level which is related to heart failure severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Free Hospital NHS Trust (RFH), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised patient data will be shared with bioengineers at Gent University in Belgium who will create the digital twins.